CLINICAL TRIAL: NCT01133834
Title: Clinical and Laboratorial Factors Associated With the Severity of Meningococcal Disease
Brief Title: Correlation Between Cytokines and the Severity of Meningococcal Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto de Infectologia Emílio Ribas (Unknown)
Responsible Party: Antonio Carlos Seguro, University of São Paulo School of Medicine
Other Study IDs: meningococcemia
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2003-02

CONDITIONS: Meningococcemia
Keywords: meningococcal disease; cytokines
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — blood sample cerebral spinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with meningococcemia: Patients with meningococcemia admitted at the Intensive Care Unit

SUMMARY:
Objectives:

Meningococcal disease (MD) is a complex catastrophic phenomenon that can converge rapidly to irreversible septic shock, myocardial dysfunction, and profound coagulopathy. During meningococcal sepsis and meningitis, a myriad of cells release cytokines within the intravascular environment and subarachnoid space. Cytokines are key molecular messengers that play key roles in orchestrating and mediating the metabolic, endocrine and coagulation responses to meningococcal infection. The aim of the present study is to determine the profile of different cytokines in serum and cerebrospinal fluid during MD, as well as relate the level of these cytokines to severity of MD.

Design:

Prospective, nonrandomized study.

Setting:

Tertiary referral intensive care unit.

Patients:

Children and adults admitted with a clinical diagnosis of MD. Interventions: Blood and cerebrospinal fluid will sample from children and adults with MD.

DETAILED DESCRIPTION:
Meningococcal disease (MD) is a complex catastrophic phenomenon that can converge rapidly to irreversible septic shock, myocardial dysfunction, and profound coagulopathy. During meningococcal sepsis and meningitis, a myriad of cells release cytokines within the intravascular environment and subarachnoid space. Cytokines are key molecular messengers that play key roles in orchestrating and mediating the metabolic, endocrine and coagulation responses to meningococcal infection. The aim of the present study is to determine the profile of different cytokines in serum and cerebrospinal fluid during MD:

IL -4; IL-6; IL-10 and interferon alfa, as well as relate the level of these cytokines to severity of MD, evaluated by occurrence of shock, acute renal failure, disseminated intravascular coagulation and survival.

Design: Prospective, nonrandomized study. Setting: Tertiary referral intensive care unit. Patients: Children and adults admitted with a clinical diagnosis of MD. Interventions: Blood and cerebrospinal fluid will sample from children and adults with MD.

Measurements and Main Results: in process Conclusions: in process

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnostic of meningococcal disease

Exclusion Criteria:

* no meningococcal disease

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted at the Intensive Care Unit of the Instituto de Infectologia Emílio Ribas
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
shock | 24 hours
  low blood pressure

SECONDARY OUTCOMES:
acute kidney injury | 3 days
  elevation of serum creatinine levels
disseminated intravascular coagulation | 24 hours
  plaquetopenia, coagulopathy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Seguro, MD, PhD, Principal Investigator — Hospital das Clínicas USP
Locations (1):
- University of São Paulo General Hospital - LIM-12 and LIM-56, São Paulo, São Paulo, Brazil